CLINICAL TRIAL: NCT06024629
Title: cOCT Versus LC-OCT for Diagnosing Basal Cell Carcinoma: a Diagnostic Cohort Study
Status: Active, not recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0086
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Basal Cell Carcinoma
Keywords: Optical coherence tomography; Line-field confocal optical coherence tomography
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with equivocal BCC lesions: Patients with equivocal BCC lesions (18+ years) who will undergo biopsy conform regular care will undergo a cOCT and LC-OCT scan.
  Interventions: Device: cOCT and LC-OCT

INTERVENTIONS:
Device: cOCT and LC-OCT — cOCT: conventional optical coherence tomography (cOCT) is an established imaging modality within dermatology that enables visualization of the architecture of the skin with a penetration depth of 1.0 - 1.5mm.
  LC-OCT: Line-field confocal optical coherence tomography (LC-OCT) is a new emerging diagnostic modality within the field of dermatology. LC-OCT enables tridimensional imaging of the skin with a cellular resolution and BCC features on LC-OCT have been described. However, the penetration depth of LC-OCT (500µm), is limited compared to the penetration depth of cOCT (1.0-1.5mm)

SUMMARY:
Basal cell carcinoma (BCC) is the most common form of cancer among the Caucasian population. Equivocal BCC lesions are usually diagnosed by means of a punch biopsy, but since the last few decades, non-invasive imaging techniques for the diagnosis of BCC gained popularity within the field of dermatology. Conventional optical coherence tomography (cOCT) is an example of a non-invasive imaging technique. Recent studies revealed that OCT assessors may achieve high diagnostic certainty and accuracy for diagnosing BCC. However, cOCT has a limited axial and lateral resolution and can therefore only visualize the gross architecture of the skin. It has been proposed that the diagnostic certainty and accuracy of cOCT could be optimized by improving the resolution. Line-field confocal optical coherence tomography (LC-OCT) is a new non-invasive imaging technique that provides tridimensional images of the skin with a cellular resolution. Although the resolution of LC-OCT is superior to cOCT, the penetration depth of LC-OCT (500µm) is limited compared to that of cOCT (1.0-1.5mm). In the proposed study, we aim to assess whether LC-OCT is superior to cOCT in terms of diagnostic accuracy for diagnosing BCC in equivocal BCC lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients (18+) with equivocal BCC lesions undergoing biopsy conform regular care

Exclusion Criteria:

* Patients unable to sign informed consent
* Patients with clinically evident BCC lesions who do not undergo biopsy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients visiting the outpatient clinic of Maastricht University Medical Center+ (MUMC+). All included patients (18+) will undergo a punch biopsie for their equivocal BCC lesion conform regular care.
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of cOCT and LC-OCT | Measured before september 1st 2024
  Diagnostic parameters such as sensitivity, specificity, PPV, NPV and DOR will be evaluated for diagnosing BCC in patients with equivocal lesions and compared between both imaging devices.

SECONDARY OUTCOMES:
Diagnostic accuracy for BCC subtyping on cOCT and LC-OCT | Measured before september 1st 2024
  Diagnostic parameter for differentiating BCC subtypes (sBCC/nBCC/iBCC) will be evaluated and compared between both imaging devices.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht UMC+, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be shared upon reasonable request